CLINICAL TRIAL: NCT05265741
Title: A Single Site, Observational, Administered to Pregnant Women at High Risk for Gestational Diabetes Mellitus
Brief Title: Gestational Diabetes Mellitus (GDM) in Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Long Island University (Other)
Collaborators: BROOKLYN INNOSEQ INC. (Unknown)
Responsible Party: Principal Investigator, Nini Fan, Principal Investigator, Long Island University
Other Study IDs: Mamome-GDM-05
Record Dates: First submitted 2022-02-23; First posted 2022-03-03 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Gestational Diabetes Mellitus; Pregnancy Complications
Keywords: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy Complications

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gut Microbiome (Fecal Sample)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ArmA_Pregnant No Gestational Diabetes Mellitus: This group is composed of pregnant women divided into 3 subgroups, one of each trimester. This arm will be required to provide 2 fecal samples. One at the start of recruitment, and one at the end of a 4-week period of the trimester.
- ArmB_Pregnant with Gestational Diabetes Mellitus: This group is composed of pregnant women divided into 3 subgroups, one of each trimester. This arm will be required to provide 2 fecal samples. One at the start of recruitment, and one at the end of a 4-week period of the trimester.
- ArmC_Non- Pregnant Control: This group is composed of non-pregnant women. This arm will be required to provide 1 or more fecal samples. It will be used as a baseline for comparison of the microbiome

SUMMARY:
The purpose of the trial is to discover and predict the development of GDM of pregnant women in their first trimester.

DETAILED DESCRIPTION:
Gestational Diabetes Mellitus (GDM) is a type of diabetes that affects pregnant women and often develops in the middle and later stages of pregnancy. GDM can lead to adverse maternal outcomes such as preeclampsia, and postpartum hemorrhage, and undesirable infant outcomes such as macrosomia and neonatal hypoglycemia. GDM also increases the risk of long-term consequences such as the development of type 2 diabetes in mothers, metabolic syndrome, and cardiovascular diseases. Gut microbiota has been shown to play a significant role in the etiology of metabolic illnesses, and recent studies have demonstrated that the gut microbiota of GDM women is altered compared to those of healthy women.

This trial aims to identify biomarkers during the first trimester (week 8-week 12) that can predict the likelihood of developing GDM while also examining potential links between GDM and gut microbiota. To achieve these objectives, the investigators have designed a trial that involves the collection of fecal samples from pregnant women for microbiome analysis at different stages of pregnancy. Although GDM is diagnosed at or after 24 weeks, the investigators will collect samples at the first, second, and third trimesters to determine if any alterations in the microbiome occur prior to symptom onset.

ELIGIBILITY:
Inclusion Criteria:

Women between the age of 18-45 Groups A and B have to be confirmed pregnant by blood test (confirmed by medical records) Subgroups A1 and B1 are pregnant women in their first trimester Subgroups A2 and B2 are pregnant women in their second trimester Subgroups A3 and B3 are pregnant women in their third trimester

Exclusion Criteria:

History of smoking or drinking during the pregnancy History of chronic diseases (cardiac, kidney, diabetes, hypertension, IBD,etc). Laxative use within 2 days prior to sample collection (The participant will be informed of the collection procedure by the recruiter and will be made aware of this requirement, we will also confirm when the first sample is taken through a phone call if for any reason the participant still made a mistake, will ask her to collect another sample to replace it) Development of any serious pregnancy complication during the participation period (e.g preeclampsia, preterm birth, miscarriage, etc) Excessive vomiting, diarrhea, or gastrointestinal symptoms for more than 5 consecutive days during the participation period. This will be confirmed through a weekly check-up call by the on-site recruiter or by Dr.Yin if the patient seeks treatment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Asian-American women who are patients of OBGYN, Dr. Xuebin Yin
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2024-02-10 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Gestational Diabetes Mellitus (GDM) Week 8 to post-delivery throughout their entire pregnancy | Up to approximately GA Week 37

SECONDARY OUTCOMES:
Global Clinical Outcome (GCO) Rank Score (GCO Rank) | Up to approximately GA Week 37; up to approximately 12 weeks post birth
Number of Participants With OGTT Oral Glucose Intolerance Test | Up to approximately GA Week 37
Number of Participants With live Birth | Up to approximately GA Week 37
Number of Participants With Preterm Birth | Up to approximately GA Week 37
Number of Participants at GA Week 24 Without an OGTT | GA Week 24-28
Gestational age at First GDM | Up to approximately GA Week 37
Gestational age at First Preeclampsia | Up to approximately GA Week 37
Gestational age at Delivery | Up to approximately GA Week 37

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Morin, PhD, Study Chair — Long Island University; Jeanmaire Molina, PhD, Principal Investigator — Long Island University; Xuebin Yin, MD, Principal Investigator — BROOKLYN INNOSEQ INC.
Locations (1):
- Long Island University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Su M, Nie Y, Shao R, Duan S, Jiang Y, Wang M, Xing Z, Sun Q, Liu X, Xu W. Diversified gut microbiota in newborns of mothers with gestational diabetes mellitus. PLoS One. 2018 Oct 17;13(10):e0205695. doi: 10.1371/journal.pone.0205695. eCollection 2018. PMID 30332459
- [Result] Hasan S, Aho V, Pereira P, Paulin L, Koivusalo SB, Auvinen P, Eriksson JG. Gut microbiome in gestational diabetes: a cross-sectional study of mothers and offspring 5 years postpartum. Acta Obstet Gynecol Scand. 2018 Jan;97(1):38-46. doi: 10.1111/aogs.13252. PMID 29077989
- [Result] Moses RG. The recurrence rate of gestational diabetes in subsequent pregnancies. Diabetes Care. 1996 Dec;19(12):1348-50. doi: 10.2337/diacare.19.12.1348. PMID 8941462
- See also: Related Info — https://microbiomejournal.biomedcentral.com/articles/10.1186/s40168-018-0472-x
- See also: Related Info — https://gut.bmj.com/content/67/9/1614